CLINICAL TRIAL: NCT03473119
Title: Acute Effects of Particulate Matter on Pulmonary Diseases: Discovery Its Chemo-signatures
Brief Title: Evaluation of Plasma Sphingosine-1-Phosphate as A Diagnostic and Prognostic Biomarkers of Community-Acquired Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: N201602089
Record Dates: First submitted 2018-03-14; First posted 2018-03-22 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-04

CONDITIONS: Pneumonia; Chronic Obstructive Pulmonary Disease; Asthma
Keywords: Sphingosine-1-phosphate
MeSH Terms: conditions — Pneumonia; Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma and Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Control: Healthy individuals
- Asthma: Asthma acute exacerbations
- Asthma with CAP: Asthma acute exacerbations with community-acquired pneumonia
- COPD: Acute exacerbations of chronic obstructive pulmonary disease
- COPD with CAP: Acute exacerbations of chronic obstructive pulmonary disease with community-acquired pneumonia
- CAP: Community-acquired pneumonia

SUMMARY:
Pneumonia is a major infectious cause of death worldwide and imposes a considerable burden on healthcare resources. Obstructive lung diseases (COPD and Asthma) are increasingly important causes of morbidity and mortality worldwide. The patients with community-acquired pneumonia (CAP), and acute exacerbations of obstructive lung diseases commonly present with similar signs and symptoms. For antibiotic use, the rapid and accurate differentiation of clinically relevant of bacterial lower respiratory tract infections from other mimics is essential. Sphingosine-1-phosphate (S1P) is a bioactive sphingolipid has both extracellular and intracellular effects in mammalian cells. S1P is involved in many physiological processes including immune responses and endothelial barrier integrity. In term of endothelial barrier integrity, S1P plays a crucial role in protecting lungs from the pulmonary leak and lung injury. Because of the involvement in lung injury, S1P would be the potential biomarker of pneumonia. Based on the above evidence, S1P plays an essential role in the pathobiology of pneumonia was hypothesized.

DETAILED DESCRIPTION:
The study was a branch of our PM2.5 observational study (Acute Effects of Particulate Matter on Pulmonary Diseases) and mainly focus on lipid biomarker for the target diseases. Lower respiratory tract infections are the most frequent infectious cause of death worldwide[1] and impose a considerable burden on healthcare resources. Despite the advancement in treatment and diagnostic technique, the overall 30-day mortality rate of community-acquired pneumonia (CAP) is as high as 12.1% for patients who aged 65 years and older admitted to hospital[2]. Obstructive lung diseases (COPD and Asthma) are increasingly important causes of morbidity and mortality worldwide. The patients with CAP, and acute exacerbations of obstructive lung diseases commonly present with similar signs and symptoms.

The use of conventional diagnostic markers, such as complete blood count (CBC) with differential and C-reactive protein is the current mainstream method for differentiating clinically relevant to bacterial lower respiratory tract infections from other mimics. However, for patients with a clinical suspicion of infection, those conventional methods have suboptimal sensitivity and specificity[3,4] The limitations often cause the ambiguity of the initiation of antibiotic treatment. As a result, unnecessary use of antibiotics adversely affects patient outcomes. Also, inappropriate antibiotic therapy increases antibiotic resistance in patients, which poses a public health problem. Current strategies to reduce antibiotic usage have included the development of biomarker-directed treatment algorithms. However, a recent study suggested that procalcitonin-guided therapy has not been effective in reducing antibiotic use[5]. Therefore, developing new biomarkers may be the answer to the problems.

Sphingosine-1-phosphate (S1P) is a bioactive sphingolipid has both extracellular and intracellular effects in mammalian cells[6-9]. S1P is synthesized by two sphingosine kinases (SphK1 and SphK 2) and degraded by S1P lyase (S1PL)[6] S1P is a ligand for five G protein-coupled receptors, S1P receptors1-5[6,7], and also acts as an intracellular second messenger[10,11]. S1P is involved in many physiological processes including immune responses and endothelial barrier integrity[12-15]. In term of endothelial barrier integrity, S1P plays a crucial role in protecting lungs from the pulmonary leak and lung injury. [16-19] Previous research suggests that S1P signaling through S1PR1 is crucial for endothelial barrier function. [20] The S1P induces actin polymerization and then results in the spreading of endothelial cells which fills intercellular gaps. Also, the S1P-signaling can stabilize the endothelial cell-cell junctions such as adherens junction and tight junction. [21-23] Both actin-dependent outward spreading of endothelial cells and cell junction stabilization enhance the endothelial barrier function. Because of the involvement in lung injury and endothelial barrier function, S1P would be the potential biomarker of pneumonia.

For the study, a case-control design was utilized for collecting clinical samples. the investigators plan to enroll 150 individuals for each targeted disease (CAP, Asthma, Asthma with CAP, COPD, and COPD with CAP) and control. Peripheral blood will be collected from the patients presenting at the emergency department (ED) of Wan Fang Hospital for an acute event of the candidate diseases. Each recruited individual will fill out a specific questionnaire, which will include lifestyle, occupation, habits, and general dietary information. The initial peripheral blood sample will be obtained in the emergency department, and if the patients were admitted, the individual's blood sample would be collected one day before a planned discharge again. The following parameters will be recorded for each participant: sex, age, body weight, body temperature, vital signs at the ED, and clinical characteristics of the disease. The laboratory testing will include baseline analyses (hematocrit, white blood count with differential, serum sodium, and chloride), ALT, AST, CRP, BUN, and creatinine. The plasma S1P will also be tested and will be measured by ELISA. The questionnaire will provide the individual's basic information of living area, occupational environment, personal habits and family history for further analysis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic obstructive pulmonary disease (COPD; ICD-9 codes 490-492, 494, 496)
* Clinical diagnosis of Asthma (ICD-9 code 493),
* Clinical diagnosis of pneumonia (ICD-9 codes 480-488).

Exclusion Criteria:

* Underage incapacity
* Pregnant women,
* Psychiatric history
* Unfamiliar with Chinese

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The individuals who have the target diseases (CAP, Asthma, Asthma with CAP COPD, and COPD with CAP) and healthy controls will be recruited at the emergency department (ED) of Wan Fang Hospital (Taipei, Taiwan). The hospital is affiliated with Taipei Medical University and is located in the metropolitan area of Taipei City, Taiwan, at Wenshan District, and has had more than 65,000 emergency visits annually.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2016-03-19 (Actual); Primary Completion 2021-03-19 (Estimated); Study Completion 2021-03-19 (Estimated)

PRIMARY OUTCOMES:
Mortality | 3 months
  3 months mortality

SECONDARY OUTCOMES:
ICU | During the hospital admission
  ICU admission
ETT | During the hospital admission
  On Tracheal tube
BiPAP | During the hospital admission
  Using Bilevel Positive Airway Pressure
Length of Stay | During the hospital admission
  length of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- The Emergency Department of Wan Fang Hospital, Taipei, Wenshan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Metersky ML, Waterer G, Nsa W, Bratzler DW. Predictors of in-hospital vs postdischarge mortality in pneumonia. Chest. 2012 Aug;142(2):476-481. doi: 10.1378/chest.11-2393. PMID 22383662
- [Background] Hausfater P. Biomarkers and infection in the emergency unit. Med Mal Infect. 2014 Apr;44(4):139-45. doi: 10.1016/j.medmal.2014.01.002. Epub 2014 Feb 17. PMID 24556451
- [Background] Mitsuma SF, Mansour MK, Dekker JP, Kim J, Rahman MZ, Tweed-Kent A, Schuetz P. Promising new assays and technologies for the diagnosis and management of infectious diseases. Clin Infect Dis. 2013 Apr;56(7):996-1002. doi: 10.1093/cid/cis1014. Epub 2012 Dec 7. PMID 23223587
- [Background] Lindenauer PK, Shieh MS, Stefan MS, Fisher KA, Haessler SD, Pekow PS, Rothberg MB, Krishnan JA, Walkey AJ. Hospital Procalcitonin Testing and Antibiotic Treatment of Patients Admitted for Chronic Obstructive Pulmonary Disease Exacerbation. Ann Am Thorac Soc. 2017 Dec;14(12):1779-1785. doi: 10.1513/AnnalsATS.201702-133OC. PMID 28795838
- [Background] Rosen H, Goetzl EJ. Sphingosine 1-phosphate and its receptors: an autocrine and paracrine network. Nat Rev Immunol. 2005 Jul;5(7):560-70. doi: 10.1038/nri1650. PMID 15999095
- [Background] Anliker B, Chun J. Cell surface receptors in lysophospholipid signaling. Semin Cell Dev Biol. 2004 Oct;15(5):457-65. doi: 10.1016/j.semcdb.2004.05.005. PMID 15271291
- [Background] Meyer zu Heringdorf D, Liliom K, Schaefer M, Danneberg K, Jaggar JH, Tigyi G, Jakobs KH. Photolysis of intracellular caged sphingosine-1-phosphate causes Ca2+ mobilization independently of G-protein-coupled receptors. FEBS Lett. 2003 Nov 20;554(3):443-9. doi: 10.1016/s0014-5793(03)01219-5. PMID 14623109
- [Background] Usatyuk PV, He D, Bindokas V, Gorshkova IA, Berdyshev EV, Garcia JG, Natarajan V. Photolysis of caged sphingosine-1-phosphate induces barrier enhancement and intracellular activation of lung endothelial cell signaling pathways. Am J Physiol Lung Cell Mol Physiol. 2011 Jun;300(6):L840-50. doi: 10.1152/ajplung.00404.2010. Epub 2011 Apr 8. PMID 21478254
- [Background] Blom T, Slotte JP, Pitson SM, Tornquist K. Enhancement of intracellular sphingosine-1-phosphate production by inositol 1,4,5-trisphosphate-evoked calcium mobilisation in HEK-293 cells: endogenous sphingosine-1-phosphate as a modulator of the calcium response. Cell Signal. 2005 Jul;17(7):827-36. doi: 10.1016/j.cellsig.2004.11.022. Epub 2005 Jan 7. PMID 15763425
- [Background] Itagaki K, Yun JK, Hengst JA, Yatani A, Hauser CJ, Spolarics Z, Deitch EA. Sphingosine 1-phosphate has dual functions in the regulation of endothelial cell permeability and Ca2+ metabolism. J Pharmacol Exp Ther. 2007 Oct;323(1):186-91. doi: 10.1124/jpet.107.121210. Epub 2007 Jul 12. PMID 17626797
- [Background] Pappu R, Schwab SR, Cornelissen I, Pereira JP, Regard JB, Xu Y, Camerer E, Zheng YW, Huang Y, Cyster JG, Coughlin SR. Promotion of lymphocyte egress into blood and lymph by distinct sources of sphingosine-1-phosphate. Science. 2007 Apr 13;316(5822):295-8. doi: 10.1126/science.1139221. Epub 2007 Mar 15. PMID 17363629
- [Background] Rivera J, Proia RL, Olivera A. The alliance of sphingosine-1-phosphate and its receptors in immunity. Nat Rev Immunol. 2008 Oct;8(10):753-63. doi: 10.1038/nri2400. PMID 18787560
- [Background] Schuchardt M, Tolle M, Prufer J, van der Giet M. Pharmacological relevance and potential of sphingosine 1-phosphate in the vascular system. Br J Pharmacol. 2011 Jul;163(6):1140-62. doi: 10.1111/j.1476-5381.2011.01260.x. PMID 21309759
- [Background] Xiong Y, Hla T. S1P control of endothelial integrity. Curr Top Microbiol Immunol. 2014;378:85-105. doi: 10.1007/978-3-319-05879-5_4. PMID 24728594
- [Background] Dudek SM, Jacobson JR, Chiang ET, Birukov KG, Wang P, Zhan X, Garcia JG. Pulmonary endothelial cell barrier enhancement by sphingosine 1-phosphate: roles for cortactin and myosin light chain kinase. J Biol Chem. 2004 Jun 4;279(23):24692-700. doi: 10.1074/jbc.M313969200. Epub 2004 Mar 31. PMID 15056655
- [Background] McVerry BJ, Peng X, Hassoun PM, Sammani S, Simon BA, Garcia JG. Sphingosine 1-phosphate reduces vascular leak in murine and canine models of acute lung injury. Am J Respir Crit Care Med. 2004 Nov 1;170(9):987-93. doi: 10.1164/rccm.200405-684OC. Epub 2004 Jul 28. PMID 15282202
- [Background] Peng X, Hassoun PM, Sammani S, McVerry BJ, Burne MJ, Rabb H, Pearse D, Tuder RM, Garcia JG. Protective effects of sphingosine 1-phosphate in murine endotoxin-induced inflammatory lung injury. Am J Respir Crit Care Med. 2004 Jun 1;169(11):1245-51. doi: 10.1164/rccm.200309-1258OC. Epub 2004 Mar 12. PMID 15020292
- [Background] Sammani S, Moreno-Vinasco L, Mirzapoiazova T, Singleton PA, Chiang ET, Evenoski CL, Wang T, Mathew B, Husain A, Moitra J, Sun X, Nunez L, Jacobson JR, Dudek SM, Natarajan V, Garcia JG. Differential effects of sphingosine 1-phosphate receptors on airway and vascular barrier function in the murine lung. Am J Respir Cell Mol Biol. 2010 Oct;43(4):394-402. doi: 10.1165/rcmb.2009-0223OC. Epub 2009 Sep 11. PMID 19749179
- [Background] Li X, Stankovic M, Bonder CS, Hahn CN, Parsons M, Pitson SM, Xia P, Proia RL, Vadas MA, Gamble JR. Basal and angiopoietin-1-mediated endothelial permeability is regulated by sphingosine kinase-1. Blood. 2008 Apr 1;111(7):3489-97. doi: 10.1182/blood-2007-05-092148. Epub 2008 Jan 16. PMID 18199826
- [Background] Camerer E, Regard JB, Cornelissen I, Srinivasan Y, Duong DN, Palmer D, Pham TH, Wong JS, Pappu R, Coughlin SR. Sphingosine-1-phosphate in the plasma compartment regulates basal and inflammation-induced vascular leak in mice. J Clin Invest. 2009 Jul;119(7):1871-9. doi: 10.1172/jci38575. PMID 19603543
- [Background] Xu M, Waters CL, Hu C, Wysolmerski RB, Vincent PA, Minnear FL. Sphingosine 1-phosphate rapidly increases endothelial barrier function independently of VE-cadherin but requires cell spreading and Rho kinase. Am J Physiol Cell Physiol. 2007 Oct;293(4):C1309-18. doi: 10.1152/ajpcell.00014.2007. Epub 2007 Aug 1. PMID 17670896
- [Background] Arce FT, Whitlock JL, Birukova AA, Birukov KG, Arnsdorf MF, Lal R, Garcia JG, Dudek SM. Regulation of the micromechanical properties of pulmonary endothelium by S1P and thrombin: role of cortactin. Biophys J. 2008 Jul;95(2):886-94. doi: 10.1529/biophysj.107.127167. Epub 2008 Apr 11. PMID 18408039